CLINICAL TRIAL: NCT06830317
Title: A Multicenter, Observational, Prospective Study on the Efficacy of Endoscopic Radiofrequency Treatment in Reducing the Need for Blood Transfusions Compared with Conventional Therapies in Patients with Gastric Antral Vascular Ectasia (GAVE)
Brief Title: Study on the Efficacy of Endoscopic Radiofrequency Treatment in Reducing the Need for Blood Transfusions in GAVE
Acronym: GAVE
Status: Not yet recruiting | Type: Observational
Sponsor: Azienda Ospedaliera Specializzata in Gastroenterologia Saverio de Bellis (Other)
Collaborators: Medtronic (Industry)
Responsible Party: Principal Investigator, Antonio Pisani, MD, Azienda Ospedaliera Specializzata in Gastroenterologia Saverio de Bellis
Other Study IDs: GAVE_STUDY
Record Dates: First submitted 2025-02-11; First posted 2025-02-17 (Actual); Last update posted 2025-02-17 (Actual); Status verified 2025-02

CONDITIONS: GAVE - Gastric Antral Vascular Ectasia
Keywords: GAVE, RADIOFREQUENCY TREATMENT, BLOOD TRANSFUSION
MeSH Terms: conditions — Gastric Antral Vascular Ectasia | interventions — Radiofrequency Ablation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- cohort: Patients with existing diagnosis of GAVE (validated by an external expert)
  Interventions: Procedure: Endoscopic Radiofrequency treatment; Other: QoL EQ5D questionaire

INTERVENTIONS:
Procedure: Endoscopic Radiofrequency treatment — Treatment with RFA will carried out with focal RFA with a TTS catheter at 12 Joule/cm2 to all visible areas of GAVE under conscious sedation or propofol sedation by experienced team of endoscopists and anesthetists
  Other Names: RFA with a TTS catheter at 12 Joule/cm2
Other: QoL EQ5D questionaire — Quality of Life EQ5D (by EuroQol Group) before every RFA treatment and at Follow up visits (3, 6 and 12 months after the first procedure). QoL questionnaire EQ5D The descriptive system comprises five dimensions: mobility, self-care, usual activities, pain/discomfort and anxiety/depression. Each dimension has 5 levels: no problems, slight problems, moderate problems, severe problems and extreme problems. The patient is asked to indicate his/her health state by ticking the box next to the most appropriate statement in each of the five dimensions. This decision results in a 1-digit number that expresses the level selected for that dimension. The digits for the five dimensions can be combined into a 5-digit number that describes the patient's health state

SUMMARY:
The aim of the study therefore is to permanently resolve the existence of the bleeding sites caused by Gave and reduce both bleeding episodes and the need for transfusion in such patients applying "Barrx" (trademark) radiofrequency endoscopic ablation technology in selected cohort of patients that will be defined the patient inclusion section.

DETAILED DESCRIPTION:
In the period from March 2025 to June 2027 n. 80 patients from 21 different medical Centers across Italy will be screened and their endoscopic findings will be shared centrally for the approval and confirmation of the GAVE diagnosis.

Formal written informed consent will take from patients to join the study. The study will be approved by our Ethics Committee of the promoting center (conforming to the 1975 Declaration of Helsinki).

Inclusion and exclusion criteria will be applied until the expected sample size is reached.

Following the GAVE diagnosis confirmation, all consecutive patients will be enrolled in the study and directed to the initial assessment before the treatment procedures. It is estimated that each center will aim to enroll n. 3-5 of pts in the participating centers over the next 24 months.

Treatment with Radiofrequency will carried out with focal Radiofrequency (RFA) with a through the scope (TTS) catheter at 12 J/cm2 to all visible areas of GAVE under conscious sedation or propofol sedation by experienced team of endoscopists and anesthetists. Prior to treatment, 2% N-acetylcysteine as a mucolytic will be applied.

All patients received pantoprazole (40 mg twice daily) and sucralfate (1 g three times per day) post-endoscopy for 4 weeks.

Following RFA procedures, all patients will return for a repeat endoscopy after 6 weeks for follow up post-treatment. In those for whom there will macroscopic GAVE present at this endoscopy, this will treated with Radiofrequency as at the initial therapy.

After 8 weeks following this, patients will return for a follow-up endoscopy during which images will captured of the gastric mucosa and will enter the follow-up phase during which Hb and ongoing transfusion/iron supplement will record at six and 12 months following the first procedure.

ELIGIBILITY:
Inclusion Criteria:

* At least 18 years of age
* Existing diagnosis of GAVE (validated by an external expert)
* Melena and/or hematemesis secondary to GAVE and/or iron deficiency anemia persisting despite systemic iron therapy or oral supplementation and/or (concentrated red globules) GRC transfusions for at least 6 months
* Negative colonoscopy (performed within 12 months prior to enrollment, exclusion of any site of bleeding)
* Able to comply with study requirements and understand and sign the informed consent form

Exclusion Criteria:

* Alternative causes for iron deficiency anemia (gastro-duodenal erosions and/or ulcerations, celiac disease, Inflammatory Bowel Disease (IBD), etc)
* Pregnancy
* Active malignancy (malignancy diagnosed in past five years or ongoing treatment)
* Anatomical malformations precluding treatment with RFA
* Blood coagulation deficit: International normalized ratio (INR)>2, Platelets (PLT) <50,000

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Participants will have demonstrated inadequate response or intolerance to existing standard-of-care treatments, such as argon plasma coagulation (APC), proton pump inhibitors (PPIs), or somatostatin analogs. This ensures the study evaluates the novel therapy in a population where current interventions have limitations. Patients who have not yet received any treatment for GAVE will also be eligible to assess the efficacy of the new therapy as a first-line option
Sampling Method: Probability Sample
Enrollment: 80 (Estimated)
Dates: Start 2025-04-02 (Estimated); Primary Completion 2027-07-02 (Estimated); Study Completion 2027-09-02 (Estimated)

PRIMARY OUTCOMES:
evaluation of sustained increase in Hemoglobin (Hgb) (at least Hgb 10.5 grams/deciliter) | 1 year from enrolling plus six months of follow-up
  compare the number of transfusions per patient pre and post treatment with the evaluation of sustained increase in Hgb (at least Hgb 10.5 g/dl) per patient six months after at least two sequential RFA treatments

SECONDARY OUTCOMES:
patient's need for transfusions and/or infusions of i.v. iron supplementation | 6 and 12 months after the end of RFA treatment
  evaluate the percentage of patients who achieve the goal of reducing the need for transfusion (respect of patient's clinical history) and/or infusions of i.v. iron supplementation.
endoscopic evaluation of GAVE remission | 1 year from enrolling plus six months of follow-up
  evaluate endoscopic partial or total regression of areas of GAVE after Radiofrequency treatment (by asking expert endoscopist to estimate the overall percentage change in GAVE).
cost-effectiveness analysis | 1 year from enrolling plus six months of follow-up
  cost-effectiveness analysis on the effects of Radiofrequency treatment in patients with GAVE.

CONTACTS AND LOCATIONS:
Overall Officials: Antonio Pisani, MD, Principal Investigator — National Institute of Gastroenterology Saverio De Bellis Research Hospital; Stefania Marangi, MD, Study Chair — National Institute of Gastroenterology Saverio De Bellis Research Hospital

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] RIDER JA, KLOTZ AP, KIRSNER JB. Gastritis with veno-capillary ectasia as a source of massive gastric hemorrhage. Gastroenterology. 1953 May;24(1):118-23. No abstract available. PMID 13052170
- [Background] Jabbari M, Cherry R, Lough JO, Daly DS, Kinnear DG, Goresky CA. Gastric antral vascular ectasia: the watermelon stomach. Gastroenterology. 1984 Nov;87(5):1165-70. PMID 6332757
- [Background] Dulai GS, Jensen DM, Kovacs TO, Gralnek IM, Jutabha R. Endoscopic treatment outcomes in watermelon stomach patients with and without portal hypertension. Endoscopy. 2004 Jan;36(1):68-72. doi: 10.1055/s-2004-814112. PMID 14722858
- [Background] Suit PF, Petras RE, Bauer TW, Petrini JL Jr. Gastric antral vascular ectasia. A histologic and morphometric study of "the watermelon stomach". Am J Surg Pathol. 1987 Oct;11(10):750-7. PMID 3499091
- [Background] Shander A, Cappellini MD, Goodnough LT. Iron overload and toxicity: the hidden risk of multiple blood transfusions. Vox Sang. 2009 Oct;97(3):185-97. doi: 10.1111/j.1423-0410.2009.01207.x. Epub 2009 Aug 3. PMID 19663936
- [Background] Fuccio L, Mussetto A, Laterza L, Eusebi LH, Bazzoli F. Diagnosis and management of gastric antral vascular ectasia. World J Gastrointest Endosc. 2013 Jan 16;5(1):6-13. doi: 10.4253/wjge.v5.i1.6. PMID 23330048
- [Background] McCarty TR, Rustagi T. Comparative Effectiveness and Safety of Radiofrequency Ablation Versus Argon Plasma Coagulation for Treatment of Gastric Antral Vascular Ectasia: A Systematic Review and Meta-Analysis. J Clin Gastroenterol. 2019 Sep;53(8):599-606. doi: 10.1097/MCG.0000000000001088. PMID 29952856
- [Background] Patel A, Patel S, Wickremesinghe PC, Vadada D. Radiofrequency ablation using Barrx(R) for the endoscopic treatment of gastric antral vascular ectasia: a series of three cases and a review of the literature on treatment options. Clin Exp Gastroenterol. 2017 Jul 10;10:113-120. doi: 10.2147/CEG.S80241. eCollection 2017. PMID 28744150
- [Background] Magee C, Lipman G, Alzoubaidi D, Everson M, Sweis R, Banks M, Graham D, Gordon C, Lovat L, Murray C, Haidry R. Radiofrequency ablation for patients with refractory symptomatic anaemia secondary to gastric antral vascular ectasia. United European Gastroenterol J. 2019 Mar;7(2):217-224. doi: 10.1177/2050640618814659. Epub 2018 Nov 15. PMID 31080606
- [Background] Hayashi S, Saeki S. Endoscopic microvascular architecture of the portale hypertensive gastric mucosa on narrow band imaging. Dig Endosc 2007; 19: 116-123.